CLINICAL TRIAL: NCT06511570
Title: A Phase 1, Open-Label Study Comparing the Safety, Tolerability, and Pharmacokinetics of Single-Dose Intravenous Sabirnetug (ACU193) and Multiple-Dose Subcutaneous Sabirnetug (ACU193) + rHuPH20 in Healthy Participants
Brief Title: A Study Comparing the Safety, Tolerability, and Pharmacokinetics of Sabirnetug IV and Sabirnetug + rHuPH20 SC in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acumen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACU193-102
Record Dates: First submitted 2024-07-08; First posted 2024-07-22 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): 12 participants receive sabirnetug by intravenous infusion
  Interventions: Drug: sabirnetug (ACU193)
- Arm 2 (Experimental): 16 participants receive sabirnetug + rHuPH20 by subcutaneous injection
  Interventions: Combination Product: Sabirnetug + rHuPH20

INTERVENTIONS:
Drug: sabirnetug (ACU193) — sabirnetug by intravenous infusion
  Arms: Arm 1
Combination Product: Sabirnetug + rHuPH20 — sabirnetug + rHuPH20 by subcutaneous injection
  Arms: Arm 2

SUMMARY:
A Study Comparing the Safety, Tolerability, and Pharmacokinetics of Sabirnetug IV and Sabirnetug + rHuPH20 SC in Healthy Participants

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily consents to participate in this study and provides written informed consent before the start of any study assessments.
2. Male and female participants ≥ 50 years of age.
3. Females must be of non-childbearing potential, defined as:

   1. Postmenopausal females must have had ≥12 months of spontaneous amenorrhea (with documented follicle-stimulating hormone (FSH) ≥40 milli international units (mIU)/mL) or
   2. Surgically sterile including those who have had a hysterectomy, bilateral oophorectomy, bilateral salpingectomy or bilateral tubal ligation at least 6 months before the first dose of the study drug.
4. Body mass index (BMI) between 18 and 32 kg/m2 (inclusive), and weighs ≥54 kg.
5. Screening vital signs (measured after participants have rested in a supine position for a minimum of 5 minutes) within the following ranges: heart rate: 40-100 beats per minute (bpm); systolic blood pressure (BP): 90-150 millimeter of mercury (mmHg); diastolic BP: 50-95 mmHg. Out-of-range vital signs may be repeated once at any time point during the study per Investigator discretion.
6. Sperm-producing males in a sexual relationship with females of childbearing potential (FOCBPs) must use adequate contraception (e.g., condom) and must not donate sperm, starting from Screening until 180 days after the last dose of the study drug (See Section 5.3).
7. Must be willing to abstain from smoking while confined at the CTU.
8. The participant is confirmed to have adequate venous access by study staff.
9. Is willing and able to remain in the CTU for the entire duration of each confinement period and return for outpatient visits.

Exclusion Criteria:

1. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the participant or the validity of the study results.
2. Shows signs/symptoms of dementia or has a parent with a known autosomal dominant mutation causing familial AD.
3. A clinically significant abnormal finding on the physical exam, medical history, clinical laboratory results or electrocardiogram (ECG), or at Screening. The Investigator may repeat clinical laboratory tests once to assess any out-of-range values for clinical significance.

   1. Participants with a value >2.5 times the upper limit of normal (ULN) or <60% the lower limit of normal (LLN) or any other value of concern per the Investigator will be excluded.
   2. QT corrected for heart rate by Fridericia's cube root formula (QTcF) interval is >460ms in females, QTcF>450ms in males and has ECG findings considered normal or not clinically significant by the Investigator or designee at Screening.
4. Suicide risk, as determined by meeting any of the following criteria:

   * Any suicide attempt or preparatory acts/behavior on the Columbia-Suicide Severity Rating Scale (C-SSRS) Baseline/Screening in the last six months.
   * Suicidal ideation in the last six months as defined by a positive response to Question 5 (Suicidal Ideation) on the C-SSRS Baseline/Screening.
   * Significant risk of suicide, as judged by the site Investigator.
5. Known allergy to biological products or known hypersensitivity to any component of sabirnetug or hyaluronidase, including excipients.
6. Use of any experimental agent within 6 months of the first dose of study drug.
7. Administration of vaccinations (e.g., SARS-CoV-2 [COVID-19], influenza) within 14 days of administration of the study drug.
8. Use of any over the counter (OTC) medication, nutritional or dietary supplements, homeopathic preparations, herbal remedies such as St. John's Wort Extract, or vitamins within 14 days before the first dose of the study drug until EOS without evaluation and approval by the Investigator.
9. Use of any prescription medication, starting from 14 days or 5 half-lives (whichever is longer) prior to the first dose of the study drug until EOS without evaluation and approval by the Investigator.
10. Blood or plasma donation within 7 days before the first dose of the study drug until EOS. Blood/plasma donations should not be made for at least 90 days after the last dose of the study drug.
11. Has any prior history of substance abuse or treatment (including alcohol) within the 2 years prior to the first study treatment administration.
12. Regular alcohol consumption >14 units per week (1 unit=½ pint beer, 25 mL of 40% spirit or a 125-mL glass of wine).
13. Has a positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates), cotinine, or alcohol.
14. Has a positive test for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) at screening or has been previously treated for hepatitis B, hepatitis C, or HIV infection.
15. Documented COVID-19 active infection or recent COVID-19 infection in the past 2 weeks.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
Estimate blood levels of sabirnetug (ACU193) | Group 1: Day 1 (predose) up to Day 43 Group 2: Day 1 (predose) up to Day 50
  Cmax (Maximum concentration, determined directly from individual concentration-time data)
Estimate time to reach maximum blood levels of sabirnetug (ACU193) | Group 1: Day 1 (predose) up to Day 43 Group 2: Day 1 (predose) up to Day 50
  Tmax (Time of the maximum concentration)
Estimate blood levels of sabirnetug (ACU193), terminal rate | Group 1: Day 1 (predose) up to Day 43 Group 2: Day 1 (predose) up to Day 50
  λz (The observed terminal rate constant; estimated by linear regression through at least three data points in the terminal phase of the log concentration-time profile)
Estimate time to reach half-life blood levels of sabirnetug (ACU193), half-life | Group 1: Day 1 (predose) up to Day 43 Group 2: Day 1 (predose) up to Day 50
  T1/2 (The observed terminal half-life)
Estimate blood levels of sabirnetug (ACU193), concentration-time | Group 1: Day 1 (predose) up to Day 43 Group 2: Day 1 (predose) up to Day 50
  AUC168h (Area under the concentration-time curve during a one-week dosing interval)
Estimate blood levels of sabirnetug (ACU193), last concentration-time | Group 1: Day 1 (predose) up to Day 43 Group 2: Day 1 (predose) up to Day 50
  AUClast (Area under the concentration-time curve from time zero to the time of the last quantifiable concentration; calculated using the linear trapezoidal rule)
Estimate blood levels of sabirnetug (ACU193), infinity concentration-time | Group 1: Day 1 (predose) up to Day 43 Group 2: Day 1 (predose) up to Day 50
  AUCinf (Area under the concentration-time curve from time zero extrapolated to infinity)
Estimate blood levels of sabirnetug (ACU193), extrapolation | Group 1: Day 1 (predose) up to Day 43 Group 2: Day 1 (predose) up to Day 50
  AUCExtrap (%)(The percentage of AUCinf based on extrapolation)
Estimate blood levels of sabirnetug (ACU193), Clast | Group 1: Day 1 (predose) up to Day 43 Group 2: Day 1 (predose) up to Day 50
  Clast (The last quantifiable concentration determined directly from individual concentration-time data)
Estimate time to reach last blood levels of sabirnetug (ACU193) | Group 1: Day 1 (predose) up to Day 43 Group 2: Day 1 (predose) up to Day 50
  Tlast (Time of the last quantifiable concentration)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Siemers, M.D., Study Director — Acumen Pharmaceuticals
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No